CLINICAL TRIAL: NCT01687907
Title: A Randomized Longitudinal Trial About the Effects of Music on Fear of Childbirth and Outcome of Delivery
Brief Title: The Effects of Music on Fear of Childbirth and Outcome of Delivery
Acronym: MUUSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Assi Sten, Principal investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18/2.9.2009, 178/13/03/03/2009
Record Dates: First submitted 2012-09-10; First posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Fear of Childbirth
Keywords: fear of childbirth; outcome of delivery; music; mother-baby relationship
MeSH Terms: interventions — Music Therapy

ARMS (4):
- Fear of childbirth, music (Active Comparator): Patients referred to the motherhood out-patient clinic because of fear of childbirth. Advised to active music listening. Followed up by weekly and monthly diaries and three questionnaires (when recruiting, just after the delivery and 6 months after the delivery).
  Interventions: Behavioral: Music
- Fear of childbirth, control (No Intervention): Patients referred to the motherhood out-patient clinic because of fear of childbirth. No intervention. Followed up by three questionnaires (when recruiting, just after the delivery and 6 months after the delivery).
- Nulliparous, music (Active Comparator): 300 nulliparous women recruited from the ultrasound screening. Advised to active music listening. Three questionnaires like the other arms, weekly and monthly diaries like the other music group. Screening questionnaires about fear of childbirth.
  Interventions: Behavioral: Music
- Nulliparous, control (No Intervention): 300 nulliparous women recruited from ultrasound screening. No intervention. 3 Questionnaires as all the other groups. Screening questionnaire about fear of childbirth.

INTERVENTIONS:
Behavioral: Music
  Arms: Fear of childbirth, music; Nulliparous, music

SUMMARY:
The aim of this trial is to find out if active music listening during pregnancy and delivery reliefs fear of childbirth, pain in delivery, need for analgesia during delivery and if there is an effect on delivery complications. Also we try to find out if there is any influence on mother-baby relationship.

DETAILED DESCRIPTION:
In Finland fear of childbirth is one of the common reasons for consultation of obstetrician and mother´s demand on elective caesarean section. Approximately 5-8% of pregnant women suffer from severe fear of childbirth, which disturbs their family-life and working and prevents normal preparation to childbirth and parenthood.

Listening or playing music is very common in all cultures. Even fetuses are able to hear and recognize music and babies are interested in voices and sounds of music.

Music therapy has been used in other purposes widely. It is known that music stimulates the synthesis of dopamine in brain and it has been shown that music has an influence on hypertensive rats, lowering their blood pressure. In human beings there has been pleasurable responses to music correlate with activity in brain. It has also been shown that music listening enhances cognitive recovery and mood after middle cerebral artery stroke.

A strong attachment between mother and infant is essential to child's normal developement. Mothers who suffer from very strong fear of childbirth often have difficulties in mother-infant relationship and pronounced risk of puerperal depression.

Many features in listening and playing music have something to do in bonding together in societies. Lullabies are good example of communication between parent and infant.

There has been some trials about music therapy and pregnancy but not systematic randomized trials about listening to music and its influence on pain experience, length of delivery or complications of delivery. Music has a relaxing influence on human beings and we assume that it has a positive influence on pregnant women also.

We try to find out if active listening to music has any influence on physical and mental wellbeing of pregnant women or is there any influence on fear of childbirth, outcome of delivery or mother-baby relationship.

Pregnant women referred to the outpatient clinic because of fear of childbirth have also normal appointments with obstetrician and/or midwife as needed and participating this trial has no influence on those appointments.

ELIGIBILITY:
Inclusion Criteria:

* fear of childbirth in arms 1 and 2,
* nulliparous in arms 3 and 4

Exclusion Criteria:

* not able to answer the questionnaires

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2009-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
spontaneous vaginal delivery | day of delivery
  delivery data collected from the patient records afterwards

SECONDARY OUTCOMES:
Delivery satisfaction | within three days after delivery (before leaving the postpartum ward)
  specific questionnaires

OTHER OUTCOMES:
early mother-infant relationship | 6 months after delivery
  specific questionnaires
mental wellbeing | during pregnancy and up to 6 months after delivery
  specific questionnaires and diaries

CONTACTS AND LOCATIONS:
Overall Officials: Terhi Saisto, MD,PhD, Study Director — Helsinki University Central Hospital; Assi Sten, MD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, HUS, Finland

REFERENCES:
- [Derived] O'Connell MA, Khashan AS, Leahy-Warren P, Stewart F, O'Neill SM. Interventions for fear of childbirth including tocophobia. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013321. doi: 10.1002/14651858.CD013321.pub2. PMID 34231203